CLINICAL TRIAL: NCT04649008
Title: Optimized Intracranial EEG Targeting in Focal Epilepsy Based Upon Neuroimaging Connectomics
Brief Title: Localizing Epileptic Networks Using MRI and iEEG
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 819126
Record Dates: First submitted 2020-11-23; First posted 2020-12-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy; Epilepsy Intractable; Epilepsy, Temporal Lobe
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy; Epilepsy, Temporal Lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epilepsy patient volunteers (Experimental): Patients recruited for the study with intractable epilepsy who are anticipated to undergo epilepsy surgery
  Interventions: Diagnostic Test: 3T Magnetic Resonance Imaging; Diagnostic Test: Intracranial electroencephalography recordings; Diagnostic Test: 7T Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: 3T Magnetic Resonance Imaging — Magnetic resonance imaging acquired at a field strength of 3 Tesla.
  Other Names: 3T MRI
Diagnostic Test: Intracranial electroencephalography recordings — Epilepsy patients may undergo implantation of intracranial electroencephalography (iEEG) electrodes for localization of epileptogenic foci, which also provide a means to record localized brain activity during memory or other tasks for research purposes.
  Other Names: Intracranial EEG recordings
Diagnostic Test: 7T Magnetic Resonance Imaging — Magnetic resonance imaging acquired at a field strength of 7 Tesla.
  Other Names: 7T MRI

SUMMARY:
Upon successful completion of this study, the investigators expect the study's contribution to be the development of noninvasive imaging biomarkers to predict IEEG functional dynamics and epilepsy surgical outcomes. Findings from the present study may inform current and new therapies to map and alter seizure spread, and pave the way for less invasive, better- targeted, patient-specific interventions with improved surgical outcomes. This research is relevant to public health because over 20 million people worldwide suffer from focal drug-resistant epilepsy and are potential candidates for cure with epilepsy surgical interventions.

DETAILED DESCRIPTION:
Despite recent advances in neuroimaging, approximately 2/3 of intractable epilepsy patients that undergo surgical evaluation continue to require intracranial EEG (IEEG), arguably the most invasive diagnostic test in medicine. Clinicians currently lack methods to quantitatively map noninvasive imaging measures of structure and function to IEEG. Specifically, there is a critical need to validate whole-brain noninvasive neuroimaging network- based biomarkers to guide precise placement of electrodes and translate noninvasive network neuroimaging to change the paradigms of clinical care. The long-term goal of this study is to predict IEEG functional dynamics and surgical outcomes using noninvasive MRI-based measures of structure and function. The investigators' overall objective, which is the next step toward attaining the study's long-term goal, is to develop open-source noninvasive imaging tools that map epileptic networks by integrating MRI and IEEG data. The central hypothesis is that noninvasive measures of structure and function relate to and can predict the intricate functional dynamics captured on IEEG. The central hypothesis will be tested in patients undergoing IEEG targeting the temporal lobe network by pursuing three specific aims: 1) To map the patient specific structural connectome to IEEG seizure onset and propagation, 2) To correlate seizure onset and propagation on IEEG with network measures derived from resting state functional MRI (rsfMRI), and 3) To integrate the structural (Aim 1) and functional (Aim 2) connectome with standard qualitative clinical data to predict IEEG network dynamics and surgical outcomes. Under the first aim patients will undergo diffusion tensor imaging (DTI) prior to stereotactic IEEG, an IEEG method that inherently samples long range networks. The functional IEEG network will be mapped to DTI thus defining how seizures are constrained by the underlying structural connectome as they propagate. Under the second aim patients with temporal lobe epilepsy will undergo rsfMRI on 7T MRI prior to stereotactic IEEG. Functional network measures from rsfMRI and IEEG will be coregistered and rsfMRI will be used to predict functional EEG ictal and interictal networks. In the third aim two models predicting IEEG network dynamics and epilepsy surgical outcomes will be created building off of methods developed in Aims 1 and 2. This research is innovative because it represents a substantive departure from the status quo by directly connecting noninvasive multimodal imaging with measures of functional network dynamics in IEEG. This research is also significant because it is expected that successful completion of these aims will yield personalized strategies for IEEG targeting based on noninvasive neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medication-refractory epilepsy
* Planned intracranial EEG (IEEG) placement
* Hypothesized to have temporal lobe epilepsy

Exclusion Criteria:

* Contraindication to 3T MRI (e.g. metal implants or claustrophobia), clinical features that typically preclude the use of IEEG (e.g. pregnancy), prior intracranial surgery or device, and IEEG findings that are non-diagnostic (e.g. seizure onset zone(s) not identified)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Structure-function coupling | Measure will be assessed upon collection of patient pre-implant MRI study and iEEG recordings, and control MRI
  This study aims to analyze MRI and iEEG to quantify structure-function coupling (SC-FC), specifically between white matter connections and IEEG, across preictal and ictal periods in consecutive patients undergoing IEEG monitoring with SEEG targeting the temporal lobe networks at the University of Pennsylvania and Medical University of South Carolina.

SECONDARY OUTCOMES:
Correlate iEEG seizure onset and propagation with 7T rsfMRI | Measure will be assessed upon collection of patient pre-implant 7T rsfMRI and iEEG recordings, and control 7T MRI
  This study aims to correlate seizure onset and propagation on IEEG with network measures derived from resting-state functional 7T MRI (rsfMRI) in MRI-negative TLE.
Imaging biomarkers for seizure onset | Measure will be assessed upon collection of patient pre-implant 3T and 7T MRI studies and iEEG recordings, and control MRI
  This study aims to correlate non-invasive structural (Outcome 1) and functional (Outcome 2) connectomes and standard clinical data with IEEG network dynamics and surgical outcomes. This represents the first quantitative multi-modal imaging study linking noninvasive imaging to IEEG functional dynamics and epilepsy surgical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Davis, MD, MSTR, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of this study and dissemination of primary study results, the analysis data files will be made available to the public, along with the final version of the study protocol, the data dictionary, and brief instructions ("Readme" file). Public use data files and the accompanying documents will be made available through the National Technical Information Service (NTIS).
  Each data file (including MRI images) will be stripped of any and all personal identifiers and will undergo de-identification. The datasets, analytical results, and analysis software used in the investigators' applications will be hosted on the NIH-funded IEEG.org portal that has been co-developed over the past almost 10 years. IEEG.org already hosts over 150 IEEG datasets and has over 3900 users, and links to software and algorithms on GitHub.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be uploaded to IEEG.org as it is collected in this study will be hosted there while funding remains available for the portal.
Access Criteria: The IEEG.org portal is open to users internationally who register or use the database as a guest.
URL: https://www.ieeg.org/

REFERENCES:
- [Background] Jette N, Wiebe S. Update on the surgical treatment of epilepsy. Curr Opin Neurol. 2013 Apr;26(2):201-7. doi: 10.1097/WCO.0b013e32835ef345. PMID 23449171
- [Background] Wiebe S. Epilepsy. Outcome patterns in epilepsy surgery--the long-term view. Nat Rev Neurol. 2012 Jan 31;8(3):123-4. doi: 10.1038/nrneurol.2012.9. PMID 22290572
- [Background] de Tisi J, Bell GS, Peacock JL, McEvoy AW, Harkness WF, Sander JW, Duncan JS. The long-term outcome of adult epilepsy surgery, patterns of seizure remission, and relapse: a cohort study. Lancet. 2011 Oct 15;378(9800):1388-95. doi: 10.1016/S0140-6736(11)60890-8. PMID 22000136
- [Background] Widdess-Walsh P, Diehl B, Najm I. Neuroimaging of focal cortical dysplasia. J Neuroimaging. 2006 Jul;16(3):185-96. doi: 10.1111/j.1552-6569.2006.00025.x. PMID 16808819
- [Background] Tassi L, Colombo N, Garbelli R, Francione S, Lo Russo G, Mai R, Cardinale F, Cossu M, Ferrario A, Galli C, Bramerio M, Citterio A, Spreafico R. Focal cortical dysplasia: neuropathological subtypes, EEG, neuroimaging and surgical outcome. Brain. 2002 Aug;125(Pt 8):1719-32. doi: 10.1093/brain/awf175. PMID 12135964
- [Background] Raybaud C, Shroff M, Rutka JT, Chuang SH. Imaging surgical epilepsy in children. Childs Nerv Syst. 2006 Aug;22(8):786-809. doi: 10.1007/s00381-006-0132-5. Epub 2006 Jul 13. PMID 16838193
- [Background] Colombo N, Tassi L, Galli C, Citterio A, Lo Russo G, Scialfa G, Spreafico R. Focal cortical dysplasias: MR imaging, histopathologic, and clinical correlations in surgically treated patients with epilepsy. AJNR Am J Neuroradiol. 2003 Apr;24(4):724-33. PMID 12695213
- [Background] Mathern GW. Challenges in the surgical treatment of epilepsy patients with cortical dysplasia. Epilepsia. 2009 Oct;50 Suppl 9:45-50. doi: 10.1111/j.1528-1167.2009.02294.x. PMID 19761453
- [Background] Wolf RL, Alsop DC, Levy-Reis I, Meyer PT, Maldjian JA, Gonzalez-Atavales J, French JA, Alavi A, Detre JA. Detection of mesial temporal lobe hypoperfusion in patients with temporal lobe epilepsy by use of arterial spin labeled perfusion MR imaging. AJNR Am J Neuroradiol. 2001 Aug;22(7):1334-41. PMID 11498422
- [Background] Detre JA, Sirven JI, Alsop DC, O'Connor MJ, French JA. Localization of subclinical ictal activity by functional magnetic resonance imaging: correlation with invasive monitoring. Ann Neurol. 1995 Oct;38(4):618-24. doi: 10.1002/ana.410380410. PMID 7574458
- [Background] Verma G, Woo JH, Chawla S, Wang S, Sheriff S, Elman LB, McCluskey LF, Grossman M, Melhem ER, Maudsley AA, Poptani H. Whole-brain analysis of amyotrophic lateral sclerosis by using echo-planar spectroscopic imaging. Radiology. 2013 Jun;267(3):851-7. doi: 10.1148/radiol.13121148. Epub 2013 Jan 29. PMID 23360740
- [Background] Maudsley AA, Domenig C, Ramsay RE, Bowen BC. Application of volumetric MR spectroscopic imaging for localization of neocortical epilepsy. Epilepsy Res. 2010 Feb;88(2-3):127-38. doi: 10.1016/j.eplepsyres.2009.10.009. Epub 2009 Nov 17. PMID 19926450
- [Background] Dlugos D, Worrell G, Davis K, Stacey W, Szaflarski J, Kanner A, Sunderam S, Rogawski M, Jackson-Ayotunde P, Loddenkemper T, Diehl B, Fureman B, Dingledine R; Epilepsy Benchmark Stewards. 2014 Epilepsy Benchmarks Area III: Improve Treatment Options for Controlling Seizures and Epilepsy-Related Conditions Without Side Effects. Epilepsy Curr. 2016 May-Jun;16(3):192-7. doi: 10.5698/1535-7511-16.3.192. No abstract available. PMID 27330452
- [Background] Khambhati AN, Davis KA, Lucas TH, Litt B, Bassett DS. Virtual Cortical Resection Reveals Push-Pull Network Control Preceding Seizure Evolution. Neuron. 2016 Sep 7;91(5):1170-1182. doi: 10.1016/j.neuron.2016.07.039. Epub 2016 Aug 25. PMID 27568515
- Available data/document: Individual Participant Data Set — https://www.ieeg.org/